CLINICAL TRIAL: NCT04375969
Title: Short to Long Effects of Whole Body Cryostimulation on Insulin Sensitivity Among Overweight: Translational Controlled Trial Investigating Coldness and Training Effects on Endocrine Regulation on Energy Metabolism
Brief Title: Short to Long Effects of Whole Body Cryostimulation on Insulin Sensitivity Among Overweight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Principal Investigator, Robert Olek, Professor, Gdansk University of Physical Education and Sport
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NCN 2017/25/B/NZ7/02309
Record Dates: First submitted 2020-04-29; First posted 2020-05-06 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Cryotherapy; Training; Overweight; Insulin
Keywords: cold treatment; insulin resistance; HIIT; cell cultures line
MeSH Terms: conditions — Overweight; Insulin Resistance | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The primary aim is to define, through a randomized controlled approach, the relative effectiveness of up to 10-20 consecutive sessions of either whole body cryostimulation (WBC), high-intensity intermittent training (HIIT), or their combination (WBC and HIIT) in improving the metabolic status of overweight subjects. The effects will be assessed, at different time-points, in terms of insulin sensitivity and modification in the profile of hormones regulating the energy metabolism (adipokines, myokines, bone-derived hormones) and the inter-organ cross-talk.
Who Masked: Participant
Masking Description: 4 groups of obese patients will take part in the study. Qualification for the test is insulin resistance, abdominal obesity, lack of physical activity, lack of cold sensitivity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- whole body cryostimulation treatment (Experimental): WBC will be performed at the Pomeranian Rheumatologic Centre in Sopot. The centre is equipped with an electric cryochamber Zimmer Medicine System, Cryochamber ELECPOL, located in a temperature- and humidity-controlled room. The patient, minimally dressed (e.g., bathing suit, socks, clogs, headband, and surgical mask), remains 30sec at -60°C (vestibule) for body adaptation and, then, passes to the cryochamber, at -110°C and stay there 3 minutes.
  Interventions: Other: whole body cryostimulation treatment
- Connection WBC treatment and HIIT training (Experimental): This group will perform HIIT protocol and WBC sessions . HIIT will be performed after 1h WBC.
  Interventions: Other: Connection WBC treatment and HIIT training
- Control Group (Active Comparator): Control group who will be investigated (meanwhile at baseline and after the interventions)
  Interventions: Other: Control Group
- HIIT training group (Experimental): This group will perform only HIIT protocol without cryo-sessions
  Interventions: Other: HIIT training group

INTERVENTIONS:
Other: whole body cryostimulation treatment — The WBC is apporved by National Ministry of Health. It uses cryochamber with low temperature -110 oC. The patient, minimally dressed (e.g., bathing suit, socks, clogs, headband, and surgical mask), remains 30sec at -60°C (vestibule) for body adaptation and, then, passes to the cryochamber, at -110°C and stay there 3 minutes.
  Arms: whole body cryostimulation treatment
Other: Connection WBC treatment and HIIT training — WBC combination with Exercise HIIT according to Litlle protocol from 2011. This exercise protocol will be applied together with cryo-sessions
  Arms: Connection WBC treatment and HIIT training
Other: Control Group — This group willnot to change their daily habits . The measurements will be taken at baseline and at the end of the study
  Arms: Control Group
Other: HIIT training group — This group will do the training program without cold exposure
  Arms: HIIT training group

SUMMARY:
Therapeutic effectiveness of coldness in relieving pain and reducing inflammation has been known for many years now. Over that time, various coldness therapies have gained in popularity, including winter swimming, snow baths or whole body cryostimulation (WBC) . Recent researches have shown positive effects of WBC on metabolic profile, low-to-moderate chronic inflammation and related diseases (e.g., obesity). WBC could be, thus, intended as an adjuvant method in the treatment of dysmetabolic conditions, such as overweight or obesity. WBC is a cheap easily accessible practice, with a few well-defined contraindications and limited non severe possible adverse events, if performed in specialized centres. At the same time, in sport science appears data, which indicated on inhibition of adaptive changes induced by regular training.

The primary aim is to define, through a randomized controlled approach, the relative effectiveness of up to 20 consecutive sessions of either WBC, high-intensity intermittent training (HIIT), or their combination (WBC and HIIT) in improving the metabolic status of overweight and obese subjects. The effects will be assessed, at different time-points, in terms of insulin sensitivity and modification in the profile of hormones regulating the energy metabolism (adipokines, myokines, bone-derived hormones) and the inter-organ cross-talk.

DETAILED DESCRIPTION:
Secondary aims are:

1. To assess the influence of WBC and HIIT on insulin sensitivity and establish the role of myokines (irisin and IL-6) in this regulation. To find the answer for the question if the rise of mentioned myokines cause a decrease of authophagy protein HMGB1.
2. To characterize potential effectiveness of these intervention protocols on bone and energy metabolisms by stimulating in vitro cultured normal human osteoblastic primary cells and β-pancreatic cells with sera obtained from patients at different time points during treatment.
3. To establish, which procedure is most effective at improving insulin sensitivity: training or training supported with WBC treatment, which factors modify this response (body composition or physical capacity of subjects)
4. To establish if training supported with WBC treatment impairs adaptive changes of trained subjects
5. To determine the potential beneficial effects of the intervention protocols on the metabolic homeostasis, and assess how long these changes are maintained over a period of four weeks or three months.

ELIGIBILITY:
Inclusion Criteria:

* obesity (BMI >30kg/m2),
* age >18 years,
* diagnosis of impaired glucose tolerance (IGT),
* functional autonomy,
* ability to discernment,
* no WBC treatment within the previous year.

Exclusion Criteria:

* using insulin or other chronic medications,
* inflammatory/immune-mediated pathologies,
* T2D,
* liver or kidney disease,
* cardiovascular diseases,
* neuropathy, retinopathy,
* neoplasia, as well as fragility fractures of bones,
* traumatic fractures in the previous 2 years,
* contraindications for WBC and exercise

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The assessment of pro- and anti-inflammatory proteins concentration in blood , in response to applied procedures. | one month
  Proinflammatory:
  HMGB1 ng/ml, CRP ng/ml TNFalpha pg/ml
  Anti-inflammaotry:
  Irisin ng/ml Adiponectin ng/ml Leptin ng/lm IL-10 pg/ml

SECONDARY OUTCOMES:
Assessment of insulin sensitivity and insulin resistance | one month
  Measurement of fasting glucose and after oral glucose test concentration:
  glucose mg/ml insulin ng/ml, calculating Matsuda and HOMA indicators based on glucose and insulin concentrations

OTHER OUTCOMES:
Expresion of proteins induced by serum collected from our subjects | 3 months
  Human osteoblasts and β-pancreatic cell line will be treated by serum, which comes from our participants
Body composition assessment | one month
  assessment of weight [kg], skeletal muscle mass [kg], fat tissue [kg]

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Ziemann, Professor, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Ziemann Ewa, Sopot, Pomeranian Voivodeship, Poland

REFERENCES:
- [Background] Lombardi G, Ziemann E, Banfi G. Whole-Body Cryotherapy in Athletes: From Therapy to Stimulation. An Updated Review of the Literature. Front Physiol. 2017 May 2;8:258. doi: 10.3389/fphys.2017.00258. eCollection 2017. PMID 28512432
- [Background] Dulian K, Laskowski R, Grzywacz T, Kujach S, Flis DJ, Smaruj M, Ziemann E. The whole body cryostimulation modifies irisin concentration and reduces inflammation in middle aged, obese men. Cryobiology. 2015 Dec;71(3):398-404. doi: 10.1016/j.cryobiol.2015.10.143. Epub 2015 Oct 22. PMID 26475491
- [Background] Ziemann E, Olek RA, Grzywacz T, Kaczor JJ, Antosiewicz J, Skrobot W, Kujach S, Laskowski R. Whole-body cryostimulation as an effective way of reducing exercise-induced inflammation and blood cholesterol in young men. Eur Cytokine Netw. 2014 Mar 1;25(1):14-23. doi: 10.1684/ecn.2014.0349. PMID 24998353